CLINICAL TRIAL: NCT02542748
Title: Comparison of Norepinephrine and Ephedrine on Hypotension After Spinal Anesthesia in Parturients Undergoing Cesarean Section: a Randomized Double Blinded Controlled Study
Brief Title: Comparison of Norepinephrine and Ephedrine on Hypotension After Spinal Anesthesia in Parturients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, Dr, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XJH-A-2015-5-5-01
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Hypotension; Obstetrical Complication of Anesthesia; Complications; Cesarean Section
Keywords: norepinephrine; ephedrine
MeSH Terms: conditions — Hypotension | interventions — Norepinephrine; Ephedrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- norepinephrine (Experimental): norepinephrine is injected after spinal anesthesia
  Interventions: Drug: Norepinephrine
- ephedrine (Other): ephedrine is injected after spinal anesthesia
  Interventions: Drug: Ephedrine

INTERVENTIONS:
Drug: Norepinephrine — norepinephrine injection
  Other Names: vasoactive agents
  Arms: norepinephrine
Drug: Ephedrine — Ephedrine injection
  Other Names: vasoactive agents
  Arms: ephedrine

SUMMARY:
Incidence of hypotension is high in parturients after spinal anesthesia. Ephedrine could be used to treat hypotension but lead to lower fetal pH as well. This study is to compare the effects of norepinephrine and ephedrine on hypotension in parturients.

DETAILED DESCRIPTION:
Spinal anesthesia is an accepted technique in elective cesarean sections. However, hypotension, resulted from sympathectomy is a common problem, especially in pregnant women. Prevention of this complication by sympathomimetic agents is of potential clinical significance. Ephedrine could be used to treat hypotension but lead to lower fetal pH, which may be related to worse fetal outcome.Norepinephrine could improve the hypotension to the same extent as phenylephrine. In this study, we tend to compare the effects of norepinephrine and ephedrine on hypotension in parturients and on fetal acid status.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective cesarean section

Exclusion Criteria:

* Patients with severe pre-eclampsia
* Patients with contraindications for spinal anesthesia
* Patients with multiple pregnancy
* Patients with gestation <38w

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
incidence of hypotension | from immediately after spinal anesthesia to 30min after spinal anesthesia

SECONDARY OUTCOMES:
pH value of fetal arterial blood | just after clamp of the umbilical cord, usually 1min to 10min after start of the surgery
incidence of nausea and vomiting | from immediately after spinal anesthesia to 30min after spinal anesthesia
incidence of dizzy | from immediately after spinal anesthesia to 30min after spinal anesthesia
incidence of chest congestion | from immediately after spinal anesthesia to 30min after spinal anesthesia
fetal arterial partial pressure of oxygen | just after clamp of the umbilical cord, usually 1min to 10min after start of the surgery
arterial base excess of fetal arterial blood | just after clamp of the umbilical cord, usually 1min to 10min after start of the surgery
lowest neonatal cerebral oxygen saturation | from clamp of the umbilical cord to 10 min later, 10min in total
lactate level of fetal arterial blood | just after clamp of the umbilical cord, usually 1min to 10min after start of the surgery
number of rescue vasoactive agent | from immediately after spinal anesthesia to 30min after spinal anesthesia
incidence of bradycardia | from immediately after spinal anesthesia to 30min after spinal anesthesia
incidence of dyspnea | from immediately after spinal anesthesia to 30min after spinal anesthesia
Apgar scores of the neonates | from clamp of umbilical cord to 1min after clamping
  The Apgar score is a method to quickly summarize the health of newborn children.It is determined by evaluating the newborn baby on five simple criteria(Appearance, Pulse, Grimace, Activity, Respiration) on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. Scores 7 and above are generally normal; 4 to 6, fairly low; and 3 and below are generally regarded as critically low and cause for immediate resuscitative efforts
Apgar scores of the neonates | from clamp of umbilical cord to 5min after clamping
  The Apgar score is a method to quickly summarize the health of newborn children.It is determined by evaluating the newborn baby on five simple criteria(Appearance, Pulse, Grimace, Activity, Respiration) on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. Scores 7 and above are generally normal; 4 to 6, fairly low; and 3 and below are generally regarded as critically low and cause for immediate resuscitative efforts

CONTACTS AND LOCATIONS:
Overall Officials: Hailong DONG, Prof., Study Chair — Xijing Hospital
Locations (1):
- Xijing Hospital,Fourth Military Medical University, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Carvalho B, Dyer RA. Norepinephrine for Spinal Hypotension during Cesarean Delivery: Another Paradigm Shift? Anesthesiology. 2015 Apr;122(4):728-30. doi: 10.1097/ALN.0000000000000602. No abstract available. PMID 25654435
- [Background] Moslemi F, Rasooli S. Comparison of Prophylactic Infusion of Phenylephrine with Ephedrine for Prevention of Hypotension in Elective Cesarean Section under Spinal Anesthesi: A Randomized Clinical Trial. Iran J Med Sci. 2015 Jan;40(1):19-26. PMID 25649721
- [Background] Mitra JK, Roy J, Bhattacharyya P, Yunus M, Lyngdoh NM. Changing trends in the management of hypotension following spinal anesthesia in cesarean section. J Postgrad Med. 2013 Apr-Jun;59(2):121-6. doi: 10.4103/0022-3859.113840. PMID 23793313
- [Derived] Fan QQ, Wang YH, Fu JW, Dong HL, Yang MP, Liu DD, Jiang XF, Wu ZX, Xiong LZ, Lu ZH. Comparison of two vasopressor protocols for preventing hypotension post-spinal anesthesia during cesarean section: a randomized controlled trial. Chin Med J (Engl). 2021 Mar 4;134(7):792-799. doi: 10.1097/CM9.0000000000001404. PMID 33661141